CLINICAL TRIAL: NCT02911454
Title: Assess the Effects of Infant Formula on Infant Stool Characteristics, Behaviour and Parental Experience in Everyday Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EBB15YE89845
Record Dates: First submitted 2016-08-30; First posted 2016-09-22 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Infant Formula

ARMS (1):
- Healthy infants: fully or partly formula fed (Experimental)
  Interventions: Other: Infant formula

INTERVENTIONS:
Other: Infant formula

SUMMARY:
A prospective, multi-country, open label study to describe the stool characteristics and behaviour as well as the parents' experience in infants receiving a recently launched infant formula in a real life situation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants, gestational age up to and including 37 weeks and 42 weeks and below. Healthy is defined as "no supervision or medical treatment by a medical specialist. Further more to be determined by HCP.
* Birth weight between 2.5 - 4.5 KG (within normal range for gestational age and sex)
* Infants up to 6 weeks of postnatal age (Including day 42)
* Receiving exclusively or at least 1 complete infant formula feeding per day at study inclusion (retrospectively exclusively or partly formula fed)
* Willingness to change from their regular infant formula to study product
* Parents' or legal guardians' aged up to and including 18 years, written, informed consent.

Exclusion Criteria:

* Infants with a congenital condition and / or previous or current illness and (or) medication that could interfere with the study
* Infants with established or suspected cows milk allergy, lactose intolerance, galactosaemia or infants on a prescribed fibre free (e.g. prebiotic oligosaccharides) diet
* Participation in any other studies involving investigational or marketed products concomitantly or within 2 weeks prior to entry into the study
* Investigator's uncertainty about the willingness of the parents / legal guardians to comply with the protocol requirements.

Ages: 1 Hour to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Stool consistency measured by Amsterdam Stool Scale. | 15 months
  Will be reported in diaries completed by the parents.
Crying time | 15 months
  Will be reported in diaries completed by the parents.
Stool frequency | 15 months
  Will be reported in diaries completed by the parents.

SECONDARY OUTCOMES:
Eating behaviour | 15 months
  Baby Eating Behaviour Questionnaire
Parental experience of child behaviour | 15 months
  PedsQL,
Impact on family life | 15 months
  FamPedsQL

CONTACTS AND LOCATIONS:
Locations (16):
- Austria (6):
  - Private practice, Bischofshofen
  - Private practice, Eferding
  - Private practice, Hallein
  - Private practice, Linz
  - Private practice, Salzburg
  - Reinhold Rauscher, Salzburg
- Poland (2):
  - Poliklinika Ginekologiczno-Poloznicza Sp. Z.O.O Sp.K, Bialystok
  - Centrum Medyczne Promed, Krakow
- Turkey (Türkiye) (8):
  - Sağlık Bilimleri Üniversitesi Ankara Eğitim ve Araştırma Hastanesi, Ankara
  - Uludağ Üniversitesi Tıp Fakültesi, Bursa
  - Haseki Eğitim ve Araştırma Hastanesi, Istanbul
  - Istanbul Florence Nightingale Hastanesi, Istanbul
  - Medipol Mega Üniversite Hastanesi, Istanbul
  - Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul
  - Sağlık Bilimleri Üniversitesi Süleymaniye Kadın Doğum ve Çocuk Hastalıkları Eğitim ve Araştırma Hastanesi, Istanbul
  - Sağlık Bilimleri Üniversitesi Ümraniye Eğitim ve Araştırma Hastanesi, Istanbul